CLINICAL TRIAL: NCT04324411
Title: Sirolimus Combined With All Trans Retinoic Acid for the Treatment of Auto-Immune Anemia
Brief Title: Sirolimus Combined With ATRA for the Treatment of Auto-Immune Anemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sirolimus-3
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Autoimmune Anemia
MeSH Terms: interventions — Sirolimus; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): combined sirolimus(serum concentration to be 4-10ng/ml) and ATRA (20mg bid) for at least 6 months
  Interventions: Drug: sirolimus and ATRA

INTERVENTIONS:
Drug: sirolimus and ATRA — sirolimus (serum concentration 4-10ng/ml) and ATRA 20mg bid

SUMMARY:
Autoimmune anemia (AIA), including autoimmune hemolytic anemia (AIHA), EVENs' syndrome (ES), acquired pure red aplastic anemia (PRCA), is a kind of anemia disease mediated by autoimmunity, which can be primary or secondary to other diseases including autoimmune disease, malignant tumor, infection, etc. Glucocorticoid is the first-line treatment. However, the recurrence rate is very high and some patients may not response to steroids, the latter defined as refractory autoimmune anemia (RAIA). Second-line therapies include cyclosporine A (CSA), cyclophosphamide, 6-mercaptopurine, CD20 monoclonal antibody, anti human lymphocyte immunoglobulin (ATG), and even splenectomy. Cyclosporine A is easy to accept while some patients may have side effects such as renal function damage, gingival hyperplasia, hypertension and so on. Other second-line drugs also have many problems, such as low effective rate, slow onset, expensive price, and large side effects, and some patients do not response to these treatments. The refractory/relapsed AIA patients have increased cardiovascular events, increased opportunities for infections, decreased quality of life, and even death. At present, there is still no effective treatment for these patients. Our previous retrospective study showed that sirolimus was effective in cyclosporine refractory PRCA with an effective rate of 70% and slight side effects. In addition, we used sirolimus in refractory AIHA and ES, with an effective rate of 60-70%. However, there are still some non-responsive patients. Recently, it has been reported that all trans retinoic acid (ATRA) combined with danazol was effective in the treatment of refractory immune thrombocytopenic purpura (ITP). Therefore, we plans to combine sirolimus and ATRA in the treatment of refractory AIA to improve the efficacy. Since both sirolimus and ATRA are cheap and have slight side effects, this combination may reduce the economic burden of patients and reduce the side effects related to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed as autoimmune anemia (autoimmune hemolytic anemia, pure red aplastic anemia, events syndrome) without organ complications;
2. ineffective, relapsed or intolerant patients who have been treated with at least one kind of sufficient current conventional drug (steroids, CsA, CD20 monoclonal antibody, tacrolimus and others) ;
3. normal cardiac function, liver function (total bilirubin ≤ 1.5 × ULN, ALT/AST ≤ 3.0 × ULN) and renal function (serum creatinine ≤ 1 × ULN);
4. no secondary disease;
5. unable to accept hematopoietic stem cell transplantation;
6. ECoG score ≤ 2;
7. able to sign the informed consent form.

Exclusion Criteria:

1. failure to make a definite diagnosis;
2. AIA secondary to known diseases such as systemic lupus erythematosus, rheumatoid arthritis, tumor or other inflammatory diseases;
3. severe hepatorenal insufficiency (creatinine, transaminase more than 3 times of the upper limit of normal value);
4. uncontrollable systemic infection or other serious diseases;
5. pregnant or lactating women;
6. patients with mental disease who are unable to sign the informed consent;
7. taking other AIA drugs or stopping the drugs for less than 3 months;
8. allergic to the study drug;
9. participation in other clinical studies;
10. patients in any other circumstances considered unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 1 year
  overall response rate
rate of side effects | 1 year
  rates and types of all side effects

SECONDARY OUTCOMES:
change of HGB concentration | through study completion, an average of 1 year
  change of HGB concentration
frequency of HGB transfusion | through study completion, an average of 1 year
  frequency of HGB transfusion
time to response | through study completion, an average of 1 year
  time to response
response duration | through study completion, an average of 1 year
  CR/PR duration
life quality score (SF 36) | through study completion, an average of 1 year
  life quality score

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: always
Access Criteria: email request